CLINICAL TRIAL: NCT02824497
Title: Early Neonatal Respiratory Distress: Changes in Level IIb Hospital Over a Period of One Year
Acronym: DROPE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DETRESSE Respiratoire
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2016-06

CONDITIONS: Neonatal Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention. It's a description study

SUMMARY:
Respiratory distress is one of the first hospital grounds during the neonatal period. The clinical presentation and severity vary by gestational age and cause. She reports to various etiological factors as maternal, neonatal or sometimes entangled. The symptomatic management has benefited from organizational progress (perinatal care) and techniques, including antenatal steroids, the use of exogenous surfactant and non-invasive ventilation early, so that the use of intubation is less frequent. The short-term evolution of patients with early respiratory distress is based on gestational age, cause and initial management.

DETAILED DESCRIPTION:
Main objective:

To describe the care and short-term respiratory become newborns 32 weeks gestation or older with early and persistent respiratory distress to 2 hours of life (H2) over a period of one year in a type IIb motherhood.

Methodology :

Design: retrospective, descriptive, single-center, non-interventional

Performed in the Saint Joseph neonatal unit. Study duration: 1 year (01/05/2013-04/30/2014).

Acquisition of data:

The patients were selected from the hospitalization reports of infants by taking the following key words: respiratory distress, invasive and noninvasive ventilation, intubation, exogenous surfactant, pneumothorax.

Data collected:

* Obstetric data:

  * Mode of delivery: route of delivery, presentation at birth.
  * Maternal morbidity.
  * antenatal corticosteroids in infants less than 34 weeks.
* Neonatal data:

  * Gestational Age
  * Birth Weight
  * cord pH
  * Apgar M5
* The terms of the allocation:

  * Tracheal Intubation
  * ventilation modes (controlled mechanical ventilation (VMC), non-invasive ventilation (NIV), nasal cannula), the maximum reached FiO2 (fraction of inspired oxygen), ventilation time for each ventilation mode. These different methods were studied in the delivery room during hospitalization (in intensive care and neonatal intensive care "NICU").
* The place of hospitalization: resuscitation and / or NICU.
* The transfer to the NICU resuscitation if necessary.
* Received drugs (exogenous surfactant, antibiotics, caffeine)
* The successful primary diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age (A) ≥ 32 SA
* Birth weight (PN) ≥ 1000 g
* Respiratory distress appeared in the first 2 of life and non-limiting in H2.

Exclusion Criteria:

* AG <32 SA
* PN <1000g
* Malformation diagnosed ante or immediate postpartum justifying a specific urgent care.
* Respiratory distress appeared before H2 and H2-limited before, whatever the company therapeutic.
* Respiratory distress appeared after H2.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants 32 weeks gestation or older with early and persistent respiratory distress to 2 hours of life (H2) over a period of one year, to a type IIb motherhood.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Obstetric data | Day 0
  Number of Participants With same characteristics for:
  * Mode of delivery: route of delivery, presentation at birth.
  * Maternal morbidity.
  * antenatal corticosteroids in infants less than 34 weeks.

SECONDARY OUTCOMES:
Neonatal data | Day 0
  Number of Participants With same characteristics for:
  * Gestational Age
  * Birth Weight
  * cord pH
  * Apgar M5
The terms of the allocation: | Day 0
  Number of Participants With same characteristics for:
  * Tracheal Intubation
  * ventilation modes (controlled mechanical ventilation (VMC), non-invasive ventilation (NIV), nasal cannula), the maximum reached FiO2, ventilation time for each ventilation mode. These different methods were studied in the delivery room during hospitalization (in intensive care and neonatal intensive care "NICU")
    * The place of hospitalization: resuscitation and / or NICU.
    * The transfer to the NICU resuscitation if necessary.
    * Received drugs (exogenous surfactant, antibiotics, caffeine)
    * The successful primary diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: WALTER Elisabeth, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France